CLINICAL TRIAL: NCT00188019
Title: Evaluation Des méthodes de dépistage du Paragangliome héréditaire Chez Les Sujets prédisposés génétiquement
Brief Title: Hereditary Paraganglioma: Evaluation of Screening Methods to Detect Tumors in SDH Positive Carriers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Collaborators: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PHRC 04-01
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2015-07-23 (Estimated); Status verified 2015-07

CONDITIONS: Paraganglioma; Pheochromocytoma
MeSH Terms: conditions — Paraganglioma; Pheochromocytoma

INTERVENTIONS:
Procedure: diagnosis methods

SUMMARY:
Hereditary paraganglioma -due to SDH (SDHD, SDHB, SDHC) germline mutations- causes paragangliomas and pheochromocytomas. Presymptomatic genetic testing should be offered to all first-degree relatives if an SDH mutation is detected in an index case with paraganglioma or pheochromocytoma. The main objective of our national clinical research project is to test different screening methods to detect presymptomatic tumors in order to establish guidelines for the work-up and the follow-up of SDH mutation carriers.

ELIGIBILITY:
Inclusion Criteria: identification of an SDH (SDHD, SDHD, SDHC) germline mutation

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 248 (Actual)
Dates: Start 2005-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vincent Rohmer, MD, Principal Investigator — University Angers Hospital; Anne-Paule Gimenez-Roqueplo, MD, PhD, Principal Investigator — Paris-Descartes University, Européen Georges Pompidou Hospital, Assistance Publique des Hôpitaux de Paris
Locations (1):
- Européen Georges Pompidou Hospital, Paris, France